CLINICAL TRIAL: NCT00951665
Title: A Phase Ib-IIa, Open-label, Dose-Escalation Study of the Safety, Tolerability and Pharmacokinetics of Trastuzumab Emtansine, Paclitaxel and Pertuzumab Administered Intravenously to Patients With Her2-positive, Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of Trastuzumab Emtansine, Paclitaxel, and Pertuzumab in Patients With HER2-Positive, Locally Advanced or Metastatic Breast Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TDM4652g; GO01355 (Other: Hoffmann-La Roche)
Record Dates: First submitted 2009-08-03; First posted 2009-08-04 (Estimated); Results first posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Metastatic Breast Cancer
Keywords: Trastuzumab DM1 (T-DM1); Trastuzumab emtansine; Armed Herceptin; HER2; HER2+; HER2 Positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Paclitaxel; pertuzumab; Ado-Trastuzumab Emtansine

ARMS (6):
- Phase lb Regimen 1 (Experimental): Participants received trastuzumab emtansine (T-DM1) every three weeks (Q3W) + paclitaxel weekly (QW) intravenously.
  Interventions: Drug: trastuzumab emtansine [Kadcyla]; Drug: paclitaxel
- Phase Ib Regimen 2 (Experimental): Participants received T-DM1 Q3W + paclitaxel QW + pertuzumab Q3W intravenously.
  Interventions: Drug: pertuzumab [Perjeta]; Drug: trastuzumab emtansine [Kadcyla]; Drug: paclitaxel
- Phase Ib Regimen 3 (Experimental): Participants received T-DM1 QW + paclitaxel QW intravenously.
  Interventions: Drug: trastuzumab emtansine [Kadcyla]; Drug: paclitaxel
- Phase Ib Regimen 4 (Experimental): Participants received T-DM1 QW + paclitaxel QW + pertuzumab Q3W intravenously.
  Interventions: Drug: pertuzumab [Perjeta]; Drug: trastuzumab emtansine [Kadcyla]; Drug: paclitaxel
- Phase IIa Group A (Experimental): Participants received maximum tolerated dose (MTD) from Phase 1b i.e. T-DM1 3.6mg/kg Q3W + paclitaxel 80mg/m^2 QW intravenously.
  Interventions: Drug: paclitaxel; Drug: trastuzumab emtansine [Kadcyla]
- Phase IIa Group B (Experimental): Participants received MTD from Phase 1b i.e. T-DM1 3.6mg/kg Q3W + paclitaxel 80mg/m^2 QW + pertuzumab Q3W intravenously.
  Interventions: Drug: paclitaxel; Drug: pertuzumab [Perjeta]; Drug: trastuzumab emtansine [Kadcyla]

INTERVENTIONS:
Drug: paclitaxel — Intravenous repeating dose
  Arms: Phase IIa Group A; Phase IIa Group B
Drug: pertuzumab [Perjeta] — Intravenous repeating dose
  Arms: Phase IIa Group B; Phase Ib Regimen 2; Phase Ib Regimen 4
Drug: trastuzumab emtansine [Kadcyla] — Intravenous escalating dose
  Arms: Phase Ib Regimen 2; Phase Ib Regimen 3; Phase Ib Regimen 4; Phase lb Regimen 1
Drug: paclitaxel — Intravenous escalating dose
  Arms: Phase Ib Regimen 2; Phase Ib Regimen 3; Phase Ib Regimen 4; Phase lb Regimen 1
Drug: trastuzumab emtansine [Kadcyla] — Intravenous repeating dose
  Arms: Phase IIa Group A; Phase IIa Group B

SUMMARY:
This Phase Ib-IIa, multi-institutional, open-label, dose-escalation study is designed to evaluate the safety, tolerability, pharmacokinetics and feasibility of trastuzumab emtansine (T-DM1) administered by intravenous (IV) infusion in combination with paclitaxel (and pertuzumab, if applicable) in patients with human epidermal growth factor receptor 2-positive (HER2-positive), locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented HER2-positive locally advanced or metastatic breast cancer
* Tumor tissue blocks or 15-20 unstained tissue slides for confirmatory central laboratory HER2 status testing and other exploratory assessments
* Prior trastuzumab in any line of therapy (Phase Ib patients only)
* No prior T-DM1 or pertuzumab therapy
* Measurable or evaluable disease
* Cardiac ejection fraction >=50% by either echocardiogram or multigated acquisition scan
* Life expectancy >= 90 days as assessed by the investigator

Exclusion Criteria:

* Fewer than 21 days since the last anti-tumor therapy, including chemotherapy, biologic, experimental, immune, hormonal or radiotherapy for the treatment of breast cancer, with the following exceptions: hormone-replacement therapy or oral contraceptives are allowed; palliative radiation therapy involving <=25% of marrow-bearing bone is allowed if completed within >= 14 days prior to first study treatment
* History of intolerance or hypersensitivity to trastuzumab and/or adverse events related to trastuzumab, murine proteins, or any of the excipients that resulted in trastuzumab being permanently discontinued
* Peripheral neuropathy of Grade >= 2 per NCI CTCAE, Version 3.0, at the time of, or within 3 weeks prior to, the first study therapy (Phase Ib patients)
* Peripheral neuropathy of Grade >/=1 per NCI CTCAE, Version 3.0, at the time of, or within 3 weeks prior to, the first study therapy (Phase IIa patients)
* History of exposure to the following cumulative doses of anthracyclines: Doxorubicin > 500 mg/m^2; Liposomal doxorubicin > 900 mg/m^2; Epirubicin > 720 mg/m^2
* History of clinically significant cardiac dysfunction
* Brain metastases that are untreated, or progressive, or have required any type of therapy (including radiation, surgery, or steroids) to control symptoms from brain metastases within 60 days prior to the first study treatment.
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, basal cell carcinoma, or synchronous or subsequent HER2-positive breast cancer or other malignancy with a similar expected curative outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-08; Primary Completion 2012-02 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (5):
- United States (5):
  - Stanford, California
  - Aurora, Colorado
  - Boston, Massachusetts
  - Detroit, Michigan
  - New York, New York

REFERENCES:
- [Derived] Krop IE, Modi S, LoRusso PM, Pegram M, Guardino E, Althaus B, Lu D, Strasak A, Elias A. Phase 1b/2a study of trastuzumab emtansine (T-DM1), paclitaxel, and pertuzumab in HER2-positive metastatic breast cancer. Breast Cancer Res. 2016 Mar 15;18(1):34. doi: 10.1186/s13058-016-0691-7. PMID 26979312

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted from 21 Jul 2009 to 04 Jun 2013 at 5 centers (4 centers for Phase Ib and 5 centers for Phase IIa) in the United States.
Groups:
- Phase Ib Regimen 1: Participants received trastuzumab emtansine (T-DM1) every three weeks (Q3W) + paclitaxel weekly (QW) intravenously.
- Phase IIa Group B: Participants received T-DM1 3.6mg/kg Q3W + paclitaxel 80mg/m^2 QW + pertuzumab Q3W intravenously.
Period: Phase 1b
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Started | 29 | 10 | 21 | 3 | 0 | 0
Started Treatment | 26 | 10 | 21 | 3 | 0 | 0
Completed | 7 | 6 | 4 | 2 | 0 | 0
Not Completed | 22 | 4 | 17 | 1 | 0 | 0
Not completed — Adverse Event | 2 | 1 | 0 | 1 | 0 | 0
Not completed — Death | 1 | 0 | 2 | 0 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Disease Progression | 13 | 2 | 14 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0 | 0
Period: Phase 2a
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Started | 0 | 0 | 0 | 0 | 22 | 22
Completed | 0 | 0 | 0 | 0 | 10 | 15
Not Completed | 0 | 0 | 0 | 0 | 12 | 7
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 1 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 2 | 0
Not completed — Disease Progression | 0 | 0 | 0 | 0 | 6 | 5

BASELINE CHARACTERISTICS:
Groups:
- Phase Ib Regimen 1: Participants received T-DM1 Q3W + paclitaxel QW intravenously.
- Phase IIa Group A: Participants received MTD from Phase 1b i.e. T-DM1 3.6mg/kg Q3W + paclitaxel 80mg/m^2 QW intravenously.
- Total: Total of all reporting groups
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B | Total
Number analyzed (Participants) | 26 | 10 | 21 | 3 | 22 | 22 | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.3 (12.3) | 51.3 (11.9) | 54.1 (8.5) | 49.3 (4.0) | 51.7 (11.8) | 55.1 (7.7) | 53.2 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 10 | 19 | 3 | 21 | 22 | 101
  Male | 0 | 0 | 2 | 0 | 1 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Any Adverse Events (AEs), Serious Adverse Events (SAEs), AEs of Grades 3/4, and Death
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered to be related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, or results in a congenital anomaly/birth defect.
Time Frame: Up to 30 days after the last dose of study treatment or study discontinuation/termination, whichever is later
Population: Safety Population: All participants who received at least a single dose of study medication were included.
Measure: Number; unit: participants
Groups:
- Phase IIa Group A: Participants received MTD from Phase 1b i.e. T-DM1 3.6mg/kg Q3W and paclitaxel 80mg/m^2 QW intravenously.
- Phase IIa Group B: Participants received MTD from Phase 1b , i.e. T-DM1 3.6mg/kg Q3W and paclitaxel 80mg/m^2 QW, plus pertuzumab Q3W intravenously.
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 26 | 10 | 21 | 3 | 22 | 22
participants
  Any AEs | 26 | 10 | 21 | 3 | 22 | 22
  Any SAEs | 7 | 5 | 7 | 2 | 6 | 6
  Death | 1 | 0 | 2 | 0 | 1 | 1
  Any AEs Grade 3 | 19 | 5 | 15 | 2 | 13 | 13
  Any AEs Grade 4 | 0 | 2 | 1 | 1 | 6 | 2
  AEs leading to T-DM1 discontinuation | 3 | 1 | 1 | 1 | 2 | 0
  AEs leading to paclitaxel discontinuation | 20 | 7 | 14 | 3 | 13 | 13
  AEs leading to pertuzumab discontinuation | NA — NA: Not applicable for this group | 1 | NA — NA: Not applicable for this group | 1 | NA — NA: Not applicable for this group | 0

2. Primary Outcome: Number of Participants With Dose Limiting Toxicity (DLT) of the Combination of T-DM1 and Paclitaxel When T-DM1 Was Administered on Either an Q3W or QW Schedule for Both With and Without Pertuzumab Treatment
Description: DLT is defined as one of the following toxicities related to study drug during Cycle 1, according to the NCI CTCAE, Version 3: Grade 3 or higher non-hematologic AEs; Grade 3 or higher elevation of serum bilirubin, hepatic transaminases, or alkaline phosphatase; Grade 4 or higher thrombocytopenia; Grade 4 or higher neutropenia; any subjectively intolerable toxicity related to T-DM1, paclitaxel, or pertuzumab; any treatment-related toxicity prohibiting the start of the second cycle of treatment and/or prompting to a dose delay or modification during the DLT observation period, such as prompting a dose reduction at Cycle 2 Day1.
Time Frame: Up to 23 days
Population: Safety Population: All participants of the dose finding part of the study (phase 1b) who received at least a single dose of study medication were included. Participants in Phase 1b (Regimen 1, Regimen 2, Regimen 3 and Regimen 4 [60 participants]) were considered for this analysis.
Measure: Number; unit: participants
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4
Number analyzed (Participants) | 26 | 10 | 21 | 3
participants | 0 | 0 | 0 | 0

3. Primary Outcome: Maximum Tolerated Dose of T-DM1 When T-DM1 (Q3W or QW) and Paclitaxel (QW) Was Administered With and Without Pertuzumab
Description: The MTD was defined as the highest dose of T-DM1 and paclitaxel at which 0 of 3 participants or 1 of 6 experienced a DLT, when T-DM1 (Q3W or QW) and paclitaxel (QW) was administered with and without pertuzumab treatment.
Time Frame: Days 1 to 21
Population: Safety Population: All participants of the dose finding part of the study (phase 1b) who received at least a single dose of study medication were included.
Measure: Number; unit: mg/kg
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4
Number analyzed (Participants) | 26 | 10 | 21 | 3
mg/kg | 3.6 | 3.6 | 2.4 | 2.4

4. Primary Outcome: Maximum Tolerated Dose of Paclitaxel When T-DM1 (Q3W or QW) and Paclitaxel (QW) Was Administered With and Without Pertuzumab
Description: The MTD was defined as the highest dose of paclitaxel at which 0 of 3 participants or 1 of 6 experienced a DLT, when paclitaxel (QW) and T-DM1 (Q3W or QW) was administered with and without pertuzumab treatment.
Time Frame: Days 1 to 21
Population: as for outcome 3
Measure: Number; unit: mg/m^2
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4
Number analyzed (Participants) | 26 | 10 | 21 | 3
mg/m^2 | 80 | 80 | 80 | 80

5. Primary Outcome: Number of Participants in Phase IIa of the Study Who Received 12 or More Paclitaxel Doses in Combination With T-DM1 and/or Pertuzumab
Description: Participants in Phase IIa received T-DM1 Q3W and paclitaxel in Group A and T-DM1, paclitaxel, and pertuzumab in Group B.
Time Frame: From Day 1 to 15 weeks
Population: Safety Population: All participants of the phase IIa part of the study who received at least a single dose of study medication and did not have disease progression in the first 12 weeks of study treatment were included.
Measure: Number; unit: participants
Groups:
- Phase IIa Group A: Participants received MTD from Phase Ib i.e. T-DM1 3.6mg/kg Q3W and paclitaxel 80mg/m^2 QW intravenously.
- Phase IIa Group B: Participants received T-DM1 3.6mg/kg Q3W, paclitaxel 80mg/m^2 QW, and pertuzumab 420 mg Q3W intravenously.
Arm/Group | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 21 | 22
participants | 11 | 11

6. Primary Outcome: Number of Participants Who Had Adverse Events That Required Dose Modification of T-DM1 or Paclitaxel
Description: Participants were assessed for toxicity prior to each dose of T-DM1 and paclitaxel; dosing occurred only if the clinical assessment and laboratory test values were acceptable. Dose modifications included dose delayed or any dose reduction. Participants in whom significant toxicities had not recovered to the treatment range defined by the dose modification guidelines at the time of their next scheduled dose, had their dose of T-DM1 and/or paclitaxel delayed or reduced for up to 21 days.
Time Frame: Up to 30 days after the last dose of study treatment or study discontinuation/termination, whichever is later
Population: Safety Population: All participants who received at least a single dose of study medication were included.
Measure: Number; unit: participants
Groups:
- Phase IIa Group B: Participants received of T-DM1 3.6mg/kg Q3W, paclitaxel 80mg/m^2 QW, and pertuzumab Q3W intravenously.
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 26 | 10 | 21 | 3 | 22 | 22
participants
  T-DM1 | 13 | 5 | 19 | 2 | 15 | 12
  Paclitaxel | 20 | 7 | 14 | 3 | 18 | 19

7. Primary Outcome: Maximum Serum Concentration (Cmax) of T-DM1 and Total Trastuzumab in Cycle 1 After Q3W Dose Regimen
Description: Cmax of serum T-DM1 and total trastuzumab (sum of conjugated and unconjugated trastuzumab) in Cycle 1 was estimated by non-compartmental analysis for Phase Ib when T-DM1 was administered Q3W.
Time Frame: Pre-dose, and 0.25 and 4 hours post-dose on Day 1; Day 8 (before paclitaxel infusion)
Population: Pharmacokinetics (PK) population included all participants from Phase Ib who received at least one dose of T-DM1 or paclitaxel with at least one post-dose concentration data point. Only participants with data available for this parameter were analyzed.
Measure: Mean (Standard Deviation); unit: microgram per millilitre (Mcg /mL)
Groups:
- Phase Ib Cohort A: Participants received 2 mg/kg T-DM1 Q3W and 65 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort B: Participants received 2 mg/kg T-DM1 Q3W and 80 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort 1: Participants received 2.4 mg/kg T-DM1 Q3W and 65 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort J: Participants received 2.4 mg/kg T-DM1 Q3W and 80 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort D: Participants received 3.0 mg/kg T-DM1 Q3W and 80 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort 3B: Participants received 3.6 mg/kg T-DM1 Q3W and 80 mg/m^2 paclitaxel QW intravenously.
Arm/Group | Phase Ib Cohort A | Phase Ib Cohort B | Phase Ib Cohort 1 | Phase Ib Cohort J | Phase Ib Cohort D | Phase Ib Cohort 3B
Number analyzed (Participants) | 2 | 6 | 8 | 3 | 3 | 3
microgram per millilitre (Mcg /mL)
  T-DM1 | 53.5 (3.1) | 44.9 (4.8) | 43.6 (16.3) | 54.6 (13.6) | 62.2 (18.9) | 76.1 (31.5)
  Total trastuzumab | 73.9 (33.4) | 61 (23.2) | 62 (15.2) | 55.2 (12.3) | 91 (45.4) | 87.4 (39.5)

8. Primary Outcome: Maximum Plasma Concentration (Cmax) of DM1 in Cycle 1 After Q3W Dose Regimen
Description: Cmax of plasma DM1 in Cycle 1 was estimated by non-compartmental analysis for Phase Ib when T-DM1 was administered Q3W.
Time Frame: Pre-dose, and 0.25 and 4 hours post-dose on Day 1; Day 8 (before paclitaxel infusion)
Population: PK population included all participants from Phase Ib who received at least one dose of T-DM1 or paclitaxel with at least one post-dose concentration data point. Only participants with data available for this parameter were analyzed.
Measure: Mean (Full Range); unit: nano gram per milliliter (ng/mL)
Arm/Group | Phase Ib Cohort B | Phase Ib Cohort 1 | Phase Ib Cohort J | Phase Ib Cohort D | Phase Ib Cohort 3B
Number analyzed (Participants) | 4 | 8 | 3 | 3 | 3
nano gram per milliliter (ng/mL) | 2.4 [2.0 to 2.7] | 3.4 [2.0 to 4.9] | 2.7 [2.6 to 2.8] | 3.2 [2.6 to 4.1] | 5.1 [3.2 to 6.3]

9. Primary Outcome: Area Under the Serum Concentration-time Curve of Total Exposure (AUC0-Day 21) of T-DM1 and Total Trastuzumab in Cycle 1 After Q3W Dose Regimen
Description: AUC0-21 for serum T-DM1 and total trastuzumab (sum of conjugated and unconjugated trastuzumab) in Cycle 1 was estimated by non-compartmental analysis for Phase Ib when T-DM1 was administered Q3W.
Time Frame: Pre- and post-dose (0.25 and 4 hours and Day 8 [before paclitaxel infusion) for Cycle 1 and pre- and post-dose (0.25 and 4 hours) for Cycle 2 (each cycle of 21 days)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day*mcg/mL
Arm/Group | Phase Ib Cohort A | Phase Ib Cohort B | Phase Ib Cohort 1 | Phase Ib Cohort J | Phase Ib Cohort D | Phase Ib Cohort 3B
Number analyzed (Participants) | 2 | 6 | 6 | 3 | 3 | 3
day*mcg/mL
  T-DM1 | 241 (57.2) | 216 (118) | 264 (77.4) | 271 (51.2) | 382 (140) | 523 (288)
  Total trastuzumab | 633 (496) | 518 (359) | 460 (308) | 401 (249) | 959 (609) | 764 (372)

10. Primary Outcome: Maximum Serum Concentration (Cmax) of T-DM1 and Total Trastuzumab in Cycle 1 After QW Dose Regimen
Description: Cmax for serum T-DM1 and total trastuzumab (sum of conjugated and unconjugated trastuzumab) in Cycle 1 was estimated by non-compartmental analysis when T-DM1 was administered QW.
Time Frame: Pre-dose, and 0.25 and 4 hours post-dose on Day 1; Day 8 (before paclitaxel infusion)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mcg/mL
Groups:
- Phase Ib Cohort 6: Participants received 1.2 mg/kg T-DM1 QW and 65 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort 7: Participants received 1.6 mg/kg T-DM1 QW and 65 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort 8: Participants received 2.0 mg/kg T-DM1 QW and 65 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort F: Participants received 2.4 mg/kg T-DM1 QW and 65 mg/m^2 paclitaxel QW intravenously.
- Phase Ib Cohort 4: Participants received 2.4 mg/kg T-DM1 QW and 80 mg/m^2 paclitaxel QW intravenously.
Arm/Group | Phase Ib Cohort 6 | Phase Ib Cohort 7 | Phase Ib Cohort 8 | Phase Ib Cohort F | Phase Ib Cohort 4
Number analyzed (Participants) | 3 | 9 | 3 | 3 | 3
mcg/mL
  T-DM1 | 24.3 (2.61) | 26 (11.2) | 39.4 (7.09) | 63.7 (8.72) | 87.8 (75.3)
  Total trastuzumab | 57.8 (31.7) | 39.9 (24.1) | 66.1 (25.2) | 97.6 (45.7) | 92.1 (69.4)

11. Primary Outcome: Maximum Plasma Concentration (Cmax) of DM1 in Cycle 1 After QW Dose Regimen
Description: Cmax for plasma DM1 in Cycle 1 was estimated by non-compartmental analysis for Phase Ib when T-DM1 was administered QW
Time Frame: Pre-dose, and 0.25 and 4 hours post-dose on Day 1, and Day 8 (before T-DM1 dose)
Population: as for outcome 8
Measure: Mean (Full Range); unit: ng/mL
Arm/Group | Phase Ib Cohort 6 | Phase Ib Cohort 7 | Phase Ib Cohort 8 | Phase Ib Cohort F | Phase Ib Cohort 4
Number analyzed (Participants) | 3 | 7 | 3 | 3 | 3
ng/mL | 1.0 [0.8 to 1.2] | 1.8 [0.8 to 2.7] | 3.0 [2.6 to 3.8] | 2.7 [2.2 to 3.2] | 4.0 [2.4 to 6.9]

12. Primary Outcome: Area Under the Serum Concentration-time Curve of Total Exposure (AUClast) of T-DM1 and Total Trastuzumab in Cycle 1 After QW Dose Regimen
Description: AUClast for serum T-DM1 and serum total trastuzumab (sum of conjugated and unconjugated trastuzumab) in Cycle 1 was estimated by non-compartmental analysis for Phase Ib when T-DM1 was administered QW
Time Frame: Pre-dose, and 0.25 and 4 hours post-dose on Day 1; Day 8 (before T-DM1 dose)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: day*µg/mL
Arm/Group | Phase Ib Cohort 6 | Phase Ib Cohort 7 | Phase Ib Cohort 8 | Phase Ib Cohort F | Phase Ib Cohort 4
Number analyzed (Participants) | 3 | 8 | 3 | 3 | 3
day*µg/mL
  T-DM1 | 84.6 (15.2) | 91.9 (41.8) | 150 (28.3) | 242 (18) | 165 (42.4)
  Total trastuzumab | 275 (170) | 149 (94.1) | 295 (121) | 460 (250) | 270 (62.2)

13. Primary Outcome: Maximum Plasma Concentration of Paclitaxel in Cycle 1 (in the Absence T-DM1) and Cycle 2 (in the Presence T-DM1)
Description: Plasma Cmax of paclitaxel (65 mg/m^2 and 80 mg/m^2) for Cycle 1 (in the absence T-DM1) and Cycle 2 (in the presence T-DM1) was estimated by non-compartmental analysis.
Time Frame: Pre-dose, and 0.25, 1, 2, 4, 6, and 24 hours post-dose for Cycle 1 and Cycle 2
Population: PK population included all participants from Phase Ib who received at least one dose of T-DM1 or paclitaxel with at least one post-dose concentration data point. "n" denotes number of participants who received the indicated study drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Phase Ib: For paclitaxel, plasma concentration-time data were available from 47 patients receiving administration of paclitaxel at QW doses of 65 and 80 mg/m^2.
Arm/Group | Phase Ib
Number analyzed (Participants) | 47
ng/mL
  65 mg, Cycle 1 (n = 29) | 1430 (53.5)
  65 mg, Cycle 2 (n = 24) | 1280 (59.8)
  80 mg, Cycle 1 (n = 18) | 1540 (64.4)
  80 mg, Cycle 2 (n = 17) | 1590 (56.7)

14. Primary Outcome: Area Under Plasma Concentration - Time Curve of Paclitaxel From Time 0 to Infinity (AUC0-inf) in Cycle 1 (in the Absence of T-DM1) and Cycle 2 (in the Presence of T-DM1)
Description: Plasma AUC0-inf of paclitaxel (65 mg/m^2 and 80 mg/m^2) was estimated by non-compartmental analysis in Cycle 1 (in the absence T-DM1) and Cycle 2 (in the presence T-DM1).
Time Frame: Pre-dose, and 0.25, 1, 2, 4, 6, and 24 hours post-dose for Cycle 1 and Cycle 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Phase Ib
Number analyzed (Participants) | 47
hr*ng/mL
  65 mg, Cycle 1 (n = 29) | 3440 (32.3)
  65 mg, Cycle 2 (n = 24) | 3520 (38)
  80 mg, Cycle 1 (n = 18) | 3890 (48)
  80 mg, Cycle 2 (n = 17) | 4220 (49.8)

15. Primary Outcome: An Elimination Half-life (t1/2) of Plasma Concentration of Paclitaxel in Cycle 1 (in the Absence of T-DM1) and Cycle 2 (in the Presence of T-DM1)
Description: Plasma t1/2 of paclitaxel (65 mg/m^2 and 80 mg/m^2) was estimated by non-compartmental analysis in Cycle 1 (in the absence T-DM1) and Cycle 2 (in the presence T-DM1).
Time Frame: Pre-dose, and 0.25, 1, 2, 4, 6, and 24 hours post-dose for Cycle 1 and Cycle 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Phase Ib
Number analyzed (Participants) | 47
hr
  65 mg, Cycle 1 (n = 29) | 9.89 (17.1)
  65 mg, Cycle 2 (n = 24) | 11.7 (25.1)
  80 mg, Cycle 1 (n = 18) | 8.94 (20)
  80 mg, Cycle 2 (n = 17) | 10.8 (30.8)

16. Primary Outcome: Plasma Clearance (CL) of Concentration of Paclitaxel in Cycle 1 (in the Absence of T-DM1) and Cycle 2 (in the Presence of T-DM1)
Description: Plasma CL of paclitaxel (65 mg/m^2 and 80 mg/m^2) was estimated by non-compartmental analysis for in Cycle 1 (in the absence T-DM1) and Cycle 2 (in the presence T-DM1).
Time Frame: Pre-dose, and 0.25, 1, 2, 4, 6, and 24 hours post-dose for Cycle 1 and Cycle 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/hr/m^2
Arm/Group | Phase Ib
Number analyzed (Participants) | 47
L/hr/m^2
  65 mg, Cycle 1 (n = 29) | 20.7 (31.1)
  65 mg, Cycle 2 (n = 24) | 21 (36.4)
  80 mg, Cycle 1 (n = 18) | 22.8 (51.1)
  80 mg, Cycle 2 (n = 17) | 23 (44.1)

17. Primary Outcome: An Apparent Volume of Distribution at Steady-state (Vss) of Plasma Concentration of Paclitaxel in Cycle 1 (in the Absence of T-DM1) and Cycle 2 (in the Presence of T-DM1)
Description: Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired blood concentration of a drug. Vss is the apparent volume of distribution at steady-state which is estimated by (D/AUC[0-inf]) X (AUMC[0-inf])/AUC[0-inf]) where D is the dose of study drug, AUMC(0-inf) is the area under the first moment curve extrapolated to infinity and AUC(0-inf) is the area under the plasma concentration-time curve from time zero to infinite time. The Vss of paclitaxel (65 mg/m2 and 80 mg/m2) is observed in Cycle 1 (in the absence of T-DM1) and Cycle 2 (in the presence of T-DM1).
Time Frame: Pre-dose, and 0.25, 1, 2, 4, 6, and 24 hours post-dose for Cycle 1 and Cycle 2
Population: as for outcome 13
Measure: Mean (Standard Deviation); unit: L/m^2
Arm/Group | Phase Ib
Number analyzed (Participants) | 47
L/m^2
  65 mg, Cycle 1 (n = 29) | 167 (56.3)
  65 mg, Cycle 2 (n = 24) | 220 (57.3)
  80 mg, Cycle 1 (n = 18) | 166 (78.9)
  80 mg, Cycle 2 (n = 17) | 196 (56.5)

18. Primary Outcome: Number of Participants With Change From Baseline in Cardiac Function
Description: Change in cardiac functions i.e., left ventricular ejection fraction (LVEF) and segmental wall abnormalities were assessed by echocardiogram or multigated acquisition scans. LVEF was assessed as change from baseline as 0 to <15%, >=15 to <25%, >=25%, and missing values.
Time Frame: Baseline (30 days prior to study dose), end of Cycle 2, and then every three cycles in Phase Ib and every four cycles in Phase IIa throughout the duration of the study (12 months) until disease progression or study discontinuation, whichever occurs first
Population: Safety Population: All participants who received at least a single dose of study medication were included.
Measure: Number; unit: participants
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 26 | 10 | 21 | 3 | 22 | 22
participants
  LVEF, increase | 8 | 3 | 5 | 0 | 5 | 4
  LVEF, 0 to <15% | 17 | 7 | 14 | 3 | 15 | 18
  LVEF, >=15 to <25% | 0 | 0 | 2 | 0 | 0 | 0
  LVEF, missing | 1 | 0 | 0 | 0 | 2 | 0
  New segmental wall abnormality | 0 | 1 | 0 | 0 | 3 | 1

19. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR)
Description: Participants with measurable disease (at least one lesion 2 centimeters [cm] or more on computed tomography (CT) scan or 1 cm or more on spiral CT scan) were considered for OR. ORR is defined as the percentage of patients with a complete response (CR)/partial response (PR) determined on two consecutive tumor assessments at least 4 weeks apart based on modified Response Evaluation Criteria in Solid Tumors, Version 1.0 (RECIST). CR defined as disappearance of all target and non-target lesions and normalization of tumor marker level. PR defined as at least 30 percent decrease in sum of the longest diameters of the target lesions taking as reference the baseline sum longest diameters.
Time Frame: Tumor assessments performed at the end of Cycle 2 and then every 2 cycles (i.e., Cycles 4, 6, 8, 10, etc. [each cycle of 21 days]) throughout the duration of the study (12 months) until disease progression or study discontinuation, whichever occurs first
Population: An efficacy population: All participants who received at least a single dose of study medication were included. Participants with measurable disease were considered for OR.
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 24 | 10 | 18 | 3 | 21 | 21
percentage of participants | 50.0 | 70.0 | 50.0 | 66.7 | 47.6 | 52.4

20. Secondary Outcome: Duration of Objective Response
Description: Duration of OR is only calculated for participants with OR and is defined as the time from the first tumor assessment that supports the participant's OR to disease progression or death.
Time Frame: as for outcome 19
Population: An efficacy population: All participants who received at least a single dose of study medication were included. Participants with OR were considered for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 12 | 7 | 9 | 2 | 10 | 11
months | 7.1 [4.2 to NA] — Not estimable due to limited follow-up. | NA [5.8 to NA] — Not estimable due to limited follow-up. | 7.0 [4.8 to NA] — Not estimable due to limited follow-up. | NA [NA to NA] — Not estimable due to limited follow-up. | NA [NA to NA] — Not estimable due to limited follow-up. | NA [NA to NA] — Not estimable due to limited follow-up.

21. Secondary Outcome: Percentage of Participants With Clinical Benefit
Description: Clinical benefit is defined as CR, PR, or stable disease (SD) of 6 months or more duration as assessed by the investigator. CR and PR are identified in previous outcome measure. SD is defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter since the treatment started. PD is defined as at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum longest diameter recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: as for outcome 19
Population: An efficacy population: All participants who received at least a single dose of study medication were included.
Measure: Number; unit: percentage of participants
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 26 | 10 | 21 | 3 | 22 | 22
percentage of participants | 65.4 | 80.0 | 61.9 | 66.7 | 54.5 | 59.1

22. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS is defined as the time from the first day of study treatment to documented disease progression or death on study i.e., death due to any cause within 30-days of last dose of study treatment, whichever occurs first.
Time Frame: as for outcome 19
Population: An efficacy population: All participants who received at least a single dose of study medication were included.
Measure: Median (Full Range); unit: months
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Number analyzed (Participants) | 26 | 10 | 21 | 3 | 22 | 22
months | 11.7 [1.3 to 13] | 11.9 [4.3 to 12.3] | 11.3 [1.7 to 12.0] | 11.0 [1.3 to 12.2] | 6.0 [0.1 to 10.0] | 6.6 [2.6 to 8.4]

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study treatment or study discontinuation/termination, whichever is later (Approximately 4 years)
Description: SAEs and other AEs were collected in the safety population, which was defined as all participants who received at least a single dose of study medication. There was one SAE that lead to death and the preferred term was not captured for it. The same SAE was captured as 'Death - unknown cause' in the below SAE table.
Arm/Group | Phase Ib Regimen 1 | Phase Ib Regimen 2 | Phase Ib Regimen 3 | Phase Ib Regimen 4 | Phase IIa Group A | Phase IIa Group B
Serious Adverse Events (participants affected / at risk) | 7/26 | 5/10 | 7/21 | 2/3 | 6/22 | 6/22
Other Adverse Events (participants affected / at risk) | 26/60 | 10/10 | 21/21 | 3/3 | 22/22 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Regimen 1 (N=26) | Phase Ib Regimen 2 (N=10) | Phase Ib Regimen 3 (N=21) | Phase Ib Regimen 4 (N=3) | Phase IIa Group A (N=22) | Phase IIa Group B (N=22)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Death - unknown cause (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thrombosis in device (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Ulcer (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1 | 1
Chills (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Device occlusion (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 2 | 2 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Device related infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Campylobacter infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Streptococcal sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Haemoglobin Decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
Haemorrhage (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase Ib Regimen 1 (N=60) | Phase Ib Regimen 2 (N=10) | Phase Ib Regimen 3 (N=21) | Phase Ib Regimen 4 (N=3) | Phase IIa Group A (N=22) | Phase IIa Group B (N=22)
Fatigue (General disorders) | 23 | 8 | 18 | 2 | 16 | 19
Mucosal Inflammation (General disorders) | 4 | 3 | 3 | 0 | 2 | 5
Oedema Peripheral (General disorders) | 4 | 2 | 3 | 0 | 4 | 0
Pyrexia (General disorders) | 2 | 1 | 7 | 0 | 2 | 3
Chills (General disorders) | 0 | 1 | 1 | 0 | 1 | 4
Chest pain (General disorders) | 0 | 1 | 1 | 0 | 1 | 2
Gait disturbance (General disorders) | 2 | 0 | 0 | 0 | 1 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 6 | 8 | 1 | 6 | 11
Rash (Skin and subcutaneous tissue disorders) | 5 | 7 | 6 | 2 | 3 | 9
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 2 | 3
Nail disorder (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 0 | 4 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0 | 1 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 4 | 1 | 4 | 5
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 6 | 1 | 6 | 1 | 2 | 7
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 2 | 1 | 3 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 6 | 9 | 2 | 5 | 11
Upper respiratory tract infection (Infections and infestations) | 8 | 2 | 4 | 1 | 2 | 3
Urinary tract infection (Infections and infestations) | 3 | 1 | 3 | 0 | 2 | 5
Cellulitis (Infections and infestations) | 2 | 2 | 2 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 3 | 0 | 0 | 0 | 1 | 0
Eye infection (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 3 | 7 | 2 | 9 | 7
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1 | 2 | 0 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 3 | 0 | 5 | 6
Joint stiffness (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 0 | 2 | 0 | 3 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0 | 2 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 1 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 7 | 1 | 8 | 0 | 5 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 3 | 7 | 1 | 3 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0 | 2 | 0 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 3 | 0
Depression (Psychiatric disorders) | 7 | 0 | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 4 | 2 | 2 | 0 | 3 | 2
Anxiety (Psychiatric disorders) | 2 | 2 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 4 | 2 | 4 | 0 | 0 | 2
Alanine aminotransferase increased (Investigations) | 2 | 1 | 2 | 0 | 0 | 0
Haemoglobin decreased (Investigations) | 2 | 0 | 1 | 0 | 1 | 1
Weight increased (Investigations) | 2 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 2 | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 1 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 1 | 1 | 0 | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 0 | 1 | 0 | 2 | 0
Hypertension (Vascular disorders) | 1 | 0 | 3 | 0 | 2 | 0
Hot flush (Vascular disorders) | 1 | 1 | 0 | 1 | 0 | 0
Lymphoedema (Vascular disorders) | 0 | 0 | 3 | 0 | 1 | 1
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 1 | 1 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 6 | 2 | 5 | 1 | 4 | 5
Neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 7 | 1 | 8 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 2 | 4 | 1 | 8 | 5
Leukopenia (Blood and lymphatic system disorders) | 3 | 1 | 1 | 0 | 1 | 0
Dry eye (Eye disorders) | 8 | 3 | 9 | 2 | 6 | 12
Vision blurred (Eye disorders) | 5 | 3 | 6 | 1 | 6 | 6
Lacrimation increased (Eye disorders) | 6 | 2 | 1 | 0 | 1 | 2
Conjunctivitis (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 1
Photophobia (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 1
Visual impairment (Eye disorders) | 1 | 1 | 1 | 0 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 22 | 8 | 18 | 3 | 20 | 19
Dysgeusia (Nervous system disorders) | 4 | 0 | 3 | 0 | 1 | 2
Headache (Nervous system disorders) | 3 | 3 | 4 | 0 | 4 | 4
Dizziness (Nervous system disorders) | 2 | 2 | 5 | 0 | 3 | 3
Paraesthesia (Nervous system disorders) | 2 | 1 | 0 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0 | 2 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 8 | 5 | 8 | 2 | 4 | 11
Nausea (Gastrointestinal disorders) | 7 | 3 | 10 | 0 | 9 | 9
Constipation (Gastrointestinal disorders) | 8 | 3 | 3 | 1 | 4 | 4
Dry mouth (Gastrointestinal disorders) | 5 | 1 | 6 | 1 | 3 | 1
Vomiting (Gastrointestinal disorders) | 4 | 2 | 4 | 0 | 5 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 0 | 2 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 3 | 2 | 2 | 0 | 1 | 3
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 2 | 0 | 1 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 1 | 2 | 0 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 3

LIMITATIONS AND CAVEATS:
Given the small sample size in the different patient subsets, no formal hypothesis testing was performed, and all statistical analyses should be considered descriptive and hypothesis-generating only.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.